CLINICAL TRIAL: NCT03344536
Title: A Phase Ib/II Study of Debio 1347 Plus Fulvestrant in Patients With FGFR-Amplified Endocrine Receptor Positive Metastatic Breast Cancer
Brief Title: A Study of Debio 1347 Plus Fulvestrant in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-379
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Results first posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: Debio 1347; Fulvestrant; 17-379
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; CH5183284

STUDY DESIGN:
Intervention Model Description: This is an open-label, single institution, phase Ib/phase II non-randomized trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- fulvestrant and Debio 1347 (Experimental): Fulvestrant will be administered according to its approved dose of 500 mg intramuscularly on days 1, 15, 29 and then every 28 days (+/-3 days) thereafter. Debio 1347 will be administered orally daily (1 cycle is 28 days) and the dose of Debio 1347 could be deescalated. The dosage in the phase 2 portion will be the MTD/RP2D determined in the phase 1b portion.
  Interventions: Drug: Fulvestrant; Drug: Debio 1347

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant will be administered according to its approved dose of 500 mg intramuscularly on days 1, 15, 29 and then every 28 days (+/-3 days) thereafter.
Drug: Debio 1347 — Debio 1347 will be administered orally daily (1 cycle is 28 days) and the dose of Debio 1347 could be deescalated.

SUMMARY:
The purpose of a phase Ib study is to find out the best or maximum tolerated dose of a medication or combination of medications. Therefore, the purpose of this study is to decide the best dose of the study drug, Debio 1347, that can be given in combination with the standard hormonal drug, fulvestrant. Debio 1347 and fulvestrant could shrink the cancer but it could also cause side effects. This study tells us about the side effects of these drugs when given in this new combination, and how often they occur.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females Age > 18 years
* Written informed consent and authorization obtained from the subject/HIPAAappointed legal representative prior to performing any protocol-related procedures including screening evaluations
* Patients with metastatic histologically or cytologically confirmed invasive breast cancer
* Female patients of postmenopausal status. with metastatic histologically or cytologically confirmed invasive breast cancer.
* Postmenopausal status will be defined as following:

  * Age ≥ 60 years
  * Age < 60 years and 12 months of amenorrhea plus follicle stimulating hormone and plasma estradiol levels within postmenopausal range by local laboratory assessment in the absence of oral contraceptive pills, hormone replacement therapy, or gonadotropin-releasing hormone (GnRH) agonist or antagonist
  * Prior bilateral oophorectomy
* Pre or perimenopausal women allowed with the addition of goserelin
* ECOG performance status 0 -1
* Tumor must be estrogen receptor and/or progesterone receptor positive ( i.e. Hormone receptor positive (HR+) and HER-2 negative as defined by the ASCO-CAP guidelines: HR+ is defined as expression of ER and/PR in ≥ 1% of cells, or HR+ by local laboratory or regional definition. HER2- is defined as a HER2 IHC score of 0 or 1+ , or an IHC score of 2+ accompanied by a negative fluorescence, chromogenic, or silver in situ hybridization test indicating the absence of HER2 gene amplification, or a HER2/CEP17 ratio of < 2.0, or local clinical guidelines.
* Tumors must have FGFR amplifications as determined by a CLIA certified laboratory. Patients with FGFR amplifications co-occurring with 11q amplification (CCND1, FGF3,4, 19 amplifications) are also eligible.
* Measurable or evaluable disease per RECIST1.1 or pure lytic or mixed lytic-blastic bone lesions
* No more than 1 prior chemotherapy regimen in the metastatic setting for the phase 2 portion. Patients in the phase 1 portion could have received any number of prior lines of therapy.
* Willing to undergo a new core or excisional biopsy from a metastatic, not previously irradiated tumor lesion during screening
* Life expectancy of greater than 3 months
* Archival Tumor (up to 10 unstained slides) will be obtained, whenever available for additional biomarker analyses
* Hematologic parameters:

  * White blood cell (WBC) count of > 3000/ul
  * Absolute neutrophil count (ANC) > 1000/ul
  * Platelets > 100,000/ul, hemoglobin > 9.0 g/dl
* Non-hematologic parameters:

  * Corrected calcium value </= 1.1 x ULN
  * Total bilirubin ≤1.5 x ULN (upper limit of normal) except subject with documented Gilbert"s syndrome (≤5 x ULN) or liver metastasis, who must have a baseline total bilirubin ≤3.0 mg/dL
  * AST and ALT ≤ 3 x ULN, unless associated with hepatobiliary metastases, in that case ≤5 x ULN
  * ALP </= 2.5 x ULN or </= 5.0 x ULN for patients with bone metastases
  * Gamma-glutamyltransferase </= 2.5 x ULN
  * Albumin >/= 2.5 g/dL
  * Phosphat </= 1.1 x ULN
  * Prothrombin time (PT) and/or prothrombin time international normalized ratio (PT-INR) and/or activated partial thromboplastin time (APTT) </= 1.3 x ULN
  * Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min on the basis of the

Cockcroft-Gault glomerular filtration rate estimation:

(140 - age) × (weight in kg) × (0.85 if female, 1.0 if male) 72 × (serum creatinine in mg/dL)

* Patients with "treated and stable" brain lesions for a duration of > 4 weeks may be enrolled.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication and agree to use effective contraception. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Prior Fulvestrant for metastatic breast cancer will be allowed for phase 1 portion but not for the phase 2 portion
* History of hypersensitivity to any of the excipients in the Debio 1347 formulation (lactose hydrate, microcrystalline cellulose, croscarmellose sodium, hydroxypropyl cellulose, sodium lauryl sulfate, and magnesium stearate).
* Other malignancies requiring active treatment in the last 6 months.
* Brain tumors and/or brain metastases unless they are asymptomatic, stable on recent imaging (not dated more than 30 days from the inclusion date), and have not required active treatment in the last 6 months.
* History and/or current evidence of endocrine alteration of calcium-phosphate homeostasis.
* History of myocardial infarction or stroke within 6 months, congestive heart failure greater than NYHA class II, unstable angina pectoris, unexplained recurrent syncope, cardiac arrhythmia requiring treatment or family history of sudden death from cardiacrelated causes.
* Baseline Frederica"s corrected QT (QTcF) interval greater than 470 msec (female) or greater than 450 msec (male), history of congenital long QT syndrome, the presence in the screening ECG of a conduction abnormality that in the opinion of the Investigator would preclude safe participation in this study.
* Concomitant use of a drug with a known risk of QTc prolongation
* Current anticoagulation therapy with therapeutic doses of warfarin (low-dose warfarin ≤ 1mg/day or low molecular-weight heparin are permitted).
* History and or current evidence of ectopic mineralisation/calcification including but not limited to the soft tissue, kidneys, intestine, myocardium and lung with the exception of calcified lymph nodes and asymptomatic coronary calcification.
* Concomitant use of high dose systemic steroids and other drugs such as calcitonin preparations, active Vitamin D3 preparations, estrogen preparations, selective estrogen receptor modulators, Vitamin K2 preparations, parathyroid hormones, phosphorus absorbers. Note, inhaled, topical steroids and low tapering doses of steroid especially in patients treated recently for brain metastases will be included.
* Corneal disease, such as bullous or band keratopathy, corneal desquamation, keratitis, corneal ulcer, or keratoconjunctivitis.
* Known infection requiring the systemic use of, for example, an antibiotic or antiviral agent.
* Known HIV, HBV or HCV infection.
* Known untreated or uncontrolled acute infection, including urinary tract infection, within 7 days of study entry.
* History of organ, bone marrow, or stem cell transplantation.
* Pregnant or lactating woman (any woman of childbearing potential who has menstruated within the year prior to enrolment will undergo pregnancy testing within 72 hours prior to receiving the first dose of study medication).
* Women of childbearing potential or men who are unwilling to use an appropriate method of contraception during the study period and for 6 months after completing treatment with Debio 1347. Oral or injectable contraceptive agents cannot be the sole method of contraception. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Poorly controlled diabetes mellitus or hypertension (e.g., systolic > 180 mmHg or diastolic > 100 mmHg).
* Inability or unwillingness to swallow oral medications.
* Clinically significant gastrointestinal abnormality that would affect the absorption of drug such as gastrointestinal dysfunction, malabsorption syndrome, major resection of the small bowel or total gastrectomy or inflammatory bowel disease.
* Uncontrolled hydropericardium.
* Chemotherapy or radiotherapy within 14 days prior to starting study treatment. In case of monoclonal antibodies/biologics, within 28 days prior to starting study treatment.
* Administration of investigational agents within 28 days prior to treatment initiation.
* Major surgery and surgery for brain metastases within 28 days prior to screening start. Of note, Intravenous port placement is not considered as a major surgery.
* Not recovered from AEs or toxicities due to previous treatments to a Grade 1 or less specified in NCI-CTCAE version 4.0 excepting, albumin (< 2.5 g/dL), AST and ALT in patients with liver metastases (> 5 × ULN) ALP in patients with bone metastases (> 5 × ULN) and alopecia.
* Prior use of a drug targeting FGF or FGFR. Patients previously treated with medications that affect FGFR signaling as a secondary target (e.g., multi-tyrosine kinase inhibitors that primarily inhibit VEGF, but to a lesser extent also affect FGFR signaling) can be considered after discussion with the Principal Investigator.
* Currently under alcohol or drug abuse rehabilitation or treatment program.
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.

Eligibility Note: Patients could have progressed on prior aromatase inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 10 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Komal Jhaveri, MD FACP, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorioal Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants received starting dose of Debio 1347 of 80mg, de-escalation cohort did not occur
Groups:
- Cohort 1: Fulvestrant and Debio 1347: Fulvestrant will be administered according to its approved dose of 500 mg intramuscularly on days 1, 15, 29 and then every 28 days (+/-3 days) thereafter. Debio 1347 will be administered orally daily (1 cycle is 28 days) and the dose of Debio 1347 could be deescalated. The dosage in the phase 2 portion will be the MTD/RP2D determined in the phase 1b portion.
  Fulvestrant: Fulvestrant will be administered according to its approved dose of 500 mg intramuscularly on days 1, 15, 29 and then every 28 days (+/-3 days) thereafter.
  Debio 1347: Debio 1347 will be administered orally daily (1 cycle is 28 days) and the dose of Debio 1347 could be deescalated.
- Cohort 2: Expansion: Expansion cohort
Period: Overall Study
Arm/Group | Cohort 1: Fulvestrant and Debio 1347 | Cohort 2: Expansion
Started | 10 | 0
Completed | 10 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants received starting dose of Debio 1347 of 80mg, de-escalation cohort did not occur
Groups:
- Cohort 2: Expansion cohort
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Fulvestrant and Debio 1347 | Cohort 2 | Total
Number analyzed (Participants) | 10 | 0 | 10
Age, Continuous [Median (Full Range); unit: years] | 56 [41 to 69] |  | 56 [41 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 |  | 10
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 10 |  | 10
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 9 |  | 9
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 |  | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Dose Limiting Toxicity
Description: Selected non-hematologic and hematologic toxicities, as measured by the NCI CTCAE Version 4.0, will be described by frequency and grade, by cycle and over all cycles, with the maximum grade over all cycles used as the summary measure per patient.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Fulvestrant and Debio 1347
Number analyzed (Participants) | 10
Participants
  Participants who experienced a dose limiting toxicity | 10
  Participants who did not experience a dose limiting toxicity | 0

2. Primary Outcome: Proportion of Patients Who Have a Best Overall Response
Description: Tumor response is based on the RECIST v.1.1.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Fulvestrant and Debio 1347
Number analyzed (Participants) | 10
Participants
  Progression of Disease | 2
  Not entered | 8

ADVERSE EVENTS:
Time Frame: 1 year
Description: All participants received starting dose of Debio 1347 of 80mg, de-escalation cohort did not occur
Arm/Group | Cohort 1: Fulvestrant and Debio 1347 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 9/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 0/10 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT03344536/Prot_SAP_000.pdf